CLINICAL TRIAL: NCT06880159
Title: Effects of Transcranial Direct Current Stimulation (tDCS) for Enhancing Cognitive Function in Children With Autism Spectrum Disorder
Brief Title: Transcranial Direct Current Stimulation in Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Yvonne Han, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20250123005
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder (ASD); Transcranial Direct Current Stimulation (tDCS); Electroencephalography
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-tDCS (Experimental): For active-tDCS condition, participants will receive stimulation on the dorsolateral prefrontal cortex with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds.
  Interventions: Device: tDCS with computerized cognitive training
- Sham-tDCS (Sham Comparator): For sham-tDCS condition, participants will receive initial stimulation with ramp up and ramp down mode for 30 seconds, eliciting a tingling sensation on the scalp then it will be discontinued.
  Interventions: Device: tDCS with computerized cognitive training

INTERVENTIONS:
Device: tDCS with computerized cognitive training — Participants will complete tDCS over 10 sessions in 2 weeks (once per day, for 10 consecutive working days), while performing the executive function training tasks. The training session will last for 20 minutes.

SUMMARY:
Background: Transcranial Direct Current Stimulation (tDCS) is a form of non-invasive brain stimulation that has aroused increased interests in the past decade. Not only that it is transient with little side-effects, and can be well-tolerated by children, it is also affordable and readily accessible, making it an appealing treatment option for autism spectrum disorder (ASD).

Objective: (1) To assess the therapeutic effects of tDCS when combined with cognitive training for 10 consecutive weekdays on improving cognitive processing in children with ASD, relative to control group receiving sham-stimulation, and (2) to evaluate the associated neural mechanisms underlying the treatment effect of tDCS on children with ASD.

Methods: To assess the therapeutic effects of tDCS, 90 adolescents with ASD (age 6-12 years) will be randomly assigned to active- (n=45), or sham- (n=45) tDCS groups. Twenty-minute sessions of tDCS stimulation to the left dorsolateral prefrontal cortex (DLPRC) will be provided on 10 consecutive weekdays, in conjunction with cognitive training exercises. Participants with a head circumference of less than 53 cm will receive 1.0 mA of stimulation, while those with a circumference of 53 cm or greater will receive 1.5 mA. EEG, fNIRS and neuropsychological tests will be administered before, immediately after, and 2 months after the series of tDCS sessions.

Hypothesis: The investigators hypothesize that children with ASD who are randomly assigned to receive a montage of prefrontal tDCS, with cathode (inhibitory) placed over left DLPFC and anode (excitatory) over right supraorbital region) will evidence greater improvement in executive function (primary outcome) than children with ASD who are randomly assigned to receive sham-tDCS.

In addition to testing the primary clinical outcome, stated above, in planned exploratory analyses, the investigators will also examine the effects of tDCS on secondary outcome measures of cognitive function, including information processing speed, working memory, inhibitory control, and cognitive flexibility; and conduct exploratory mediation analyses to better understand the potential neurophysiological factors underlying the therapeutic effects of tDCS. This will include E/I ratio as exploratory mediator variables. As these secondary analyses are exploratory, the investigators will report them as such in presentations and published papers, and the investigators will not draw definitive conclusions from them. Rather, they will be used to better understand the potential impact of tDCS and the mechanisms underlying impact, and to inform future research.

ELIGIBILITY:
Inclusion Criteria:

* being 8-12 years old
* diagnosed with ASD given by registered psychiatrists or clinical psychologists according to the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) criteria of ASD
* IQ score above 60
* able to communicate in Chinese

Exclusion Criteria:

* with severe motor dysfunctions
* history of other neurological and psychiatric disorders or head trauma

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Average standardised score of executive function tests | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  The executive function of the children with ASD will be assessed using the Executive Composite score, which will be derived by summing the scores from the test battery of executive functions.
  Simple-task processing speed will be evaluated using the CANTAB® 5-choice Reaction Time (RTI) task. Complex-task processing speed will be assessed using the computerized version of the Wisconsin Card Sorting Test (WCST). The mean reaction time is calculated for the trials giving a correct answer during WCST.
  The reaction time measured from both tasks will be converted to standard scores and averaged to yield an executive composite score. Lower scores indicate poorer executive functioning.

SECONDARY OUTCOMES:
Change in CANTAB® cognitive test - Reaction Time (RTI) | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  RTI assesses motor and mental response speeds, reaction time, response accuracy and impulsivity. It consists of 30 trials with five potential targets and requires participants to make flexible responses as fast as possible to the target stimulus (shown in yellow). Specifically, movement and reaction time will be measured, where shorter duration reflects faster processing speed.
Change in CANTAB® cognitive test - Stop Signal Task (SST) | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  SST assesses the ability of inhibition control. The participant must respond to an arrow stimulus, by selecting one of two options, depending on the direction in which the arrow points. If an audio tone is present, the subject must withhold making that response (inhibition). Accuracy will be measured, where higher accuracy indicates better inhibition control.
Change in CANTAB® cognitive test - Multitasking Test (MTT): Response Latencies | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  MTT assesses the ability to resolve the interference of task-irrelevant information (stroop-like effect). The test displays an arrow which can appear on either the left or right side of the screen and can point to either the left or right side. In each trial, participants are presented with a cue that indicates which button to press according to two different rules. And the rules that participants have to follow may change from trial to trial in a randomized order. Participant's response latencies will be measured.
Change in CANTAB® cognitive test - Multitasking Test (MTT): Error Scores | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  MTT assesses the ability to resolve the interference of task-irrelevant information (stroop-like effect). The test displays an arrow which can appear on either the left or right side of the screen and can point to either the left or right side. In each trial, participants are presented with a cue that indicates which button to press according to two different rules. And the rules that participants have to follow may change from trial to trial in a randomized order. Participant's error scores will be measured.
Change in CANTAB® cognitive test - Emotion Recognition Task (ERT) | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  ERT assesses ability to identify six basic emotions in facial expressions along a continuum of expression magnitude. The participants must select which emotion the facial image displayed 0.2s ago. Accuracy and its percentage, as well as response latencies will be measured.
Change in Verbal Fluency Test (VFT) | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  The VFT assesses an individual's ability of working memory retrieval and executive control by instructing the individual to generate words for given semantic categories within a limited time. The VFT experimental paradigm is designed and presented with E-prime 3 (Psychology Software Tools Inc., Sharpsburg, PA, USA). During the experimental blocks, which will be counterbalanced across individuals to avoid order effects, a category word (i.e. 'transportation' or 'country') will be shown on the screen. Participants will be asked to focus their eye gaze on the center of the screen and continuously repeat '1, 2, 3, 4' slowly during the given period of time. Their responses will be recorded by an audio recorder and then transferred into written form on an Excel spreadsheet. The number of unique and correct words generated will be counted for each of the participants. This test will be paired with fNIRS recording.

OTHER OUTCOMES:
Exploratory mediator - excitability-inhibitory (E/I) ratio (indexed by EEG measures) | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  EEG resting-state theta coherence (4-7.5 Hz) will be computed from EEG signals collected from the 19 electrode positions collected from 5-min eye opened resting. Raw data will be processed with the EEGLAB Toolbox using MATLAB® R2019a. Automatic channel rejection, re-referencing, finite impulse response filtering will be performed. To filter artifacts, visual inspection of the EEG data will also be performed. Independent component analysis (ICA) will be used to further remove muscle and eyeblink artifacts. The E/I ratio will be calculated using the method described by Bruining et al (2020). the correlation between amplitude and fluctuation will be calculated for each EEG channel to yield the E/I ratio.
Oxyhemoglobin Concentration (measured by fNIRS) | First day of intervention, 1 day and 2 months after the last day of intervention (3 time points, up to 2 months)
  fNIRS data will be collected from 15 channel positions and processed using the NIRSIT Lite Analysis Tool version 3.1.0 (OBELAB Inc., Seoul, Korea), which is a MATLAB® R2019a compatible graphical user interface. The raw light intensity data for resting-state and task-based recordings (i.e. VFT) will be converted into changes in oxyhemoglobin (oxy-Hb) concentration according to the modified Beer-Lambert Law. To remove the physiological noise and movement artifacts, a 0.005-0.05 Hz bandpass filter will be used. To avoid the contamination of data caused by head movements, which are observed as spikes or significant shifts from baseline values, two additional channel rejection measures will be taken. Baseline corrections will be performed for task-based recordings based on the mean pretask baseline values defined by 5s prior to the task blocks to control for task-irrelevant [oxy-Hb] changes. The block average fNIRS data will be used for subsequent statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Han, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong